CLINICAL TRIAL: NCT01734278
Title: An Observational Post-Authorisation Safety Specialist Cohort Monitoring Study (SCEM) to Monitor the Safety and Utilisation of Asenapine (Sycrest) in the Mental Health Trust Setting in England
Brief Title: Observational Post-Authorisation Safety Study of Asenapine (Sycrest)
Acronym: OBSERVA
Status: Completed | Type: Observational
Sponsor: Professor Saad Shakir (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Professor Saad Shakir, Director, Drug Safety Research Unit, Southampton, UK
Organization: Drug Safety Research Unit, Southampton, UK (Other)
Other Study IDs: OBSERVA
Record Dates: First submitted 2012-11-22; First posted 2012-11-27 (Estimated); Last update posted 2018-07-31 (Actual); Status verified 2018-07

CONDITIONS: Manic Disorder
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Asenapine: Patients prescribed asenapine for any indication.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — This is a non-interventional study.

SUMMARY:
The purpose of this observational study is to evaluate the use and short term safety of Asenapine (Sycrest) in real-life usage in the Mental Health Trust Setting in the United Kingdom(UK) National Health Service (NHS). The study is to be carried out independently by the Drug Safety Research Unit (DSRU) in Southampton, although it is funded by Merck, the manufacturer of Sycrest.

ELIGIBILITY:
Inclusion Criteria:

* Patients for whom a study questionnaire containing useful information has been returned

Exclusion Criteria:

* Patients who do not provide consent
* Patients within selected institutions (for example prisons)
* Patients who commenced treatment between date of market launch (to be confirmed) and study start
* Enrolled patients for whom both the baseline and 12-week questionnaires are returned blank (contain no clinical information)
* Enrolled patients for whom the psychiatrist, designated member of clinical care team, or study facilitator from the DSRU reports that the patient did not take or was never prescribed asenapine
* Enrolled patients for whom there is evidence to suggest duplication of patients
* Enrolled patients for whom informed written or verbal notification is received by DSRU indicating that they no longer wish to participate at any stage of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients prescribed asenapine in a NHS Mental Health Trust in England.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2012-10; Primary Completion 2017-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
The incidence of selected identified risks of asenapine in the mental health care trust setting | 12 weeks after asenapine is first prescribed

CONTACTS AND LOCATIONS:
Locations (1):
- South Staffordshire and Shropshire Healthcare NHS Foundation Trust, Stafford, Staffordshire, United Kingdom